CLINICAL TRIAL: NCT05417373
Title: Development and Validation of a Radiomics-based Diagnosis Model for Pulmonary Arterial Hypertension
Brief Title: Algorithms to Diagnose Pulmonary Arterial Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Xinqiao Hospital of Chongqing (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Sponsor
Other Study IDs: diagnosis of PAH
Record Dates: First submitted 2022-06-06; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Diagnosis Model; Prediction Algorithm
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The development cohort: The development cohort was composed of patients diagnosed with PAH and healthy control group from 2019.1-2021.5 in RenjiH.
- The validation cohort: The validation cohort was composed of patients are suspected as PAH by echocardiography in 2021.5-2021.12 or suspected patients are form other medical institutions.
  Interventions: Other: calculated radscore

INTERVENTIONS:
Other: calculated radscore — The development cohort is case_control research. The validation cohort is prospective study to test the accuracy of calculated radscore based on diagonisis model.
  Groups: The validation cohort

SUMMARY:
The investigators intend to evalute the value of radiomics signature of pulmonary vessels from chest computed tomography (CT) for dianosis and prognosis of pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a heterogeneous disorder composed of varying pathobiology that may involve multiple clinical conditions. Computed tomography (CT) is a minimally invasive imaging technique capable of providing both high contrast and high resolution detail of the lungs and arteries. Application of radiomics as prognosis and diagnosis tools could quantifies high-dimensional features from CT data to investigate vescualr heterogeneity.Development and validation of PAH diagnosis Algorithms based on radiomics may serve as a complementary readout to current CT-based metrics and provide valuable evidence to make the treatment management decision in early PAH.

ELIGIBILITY:
Inclusion Criteria:

1. Chest CT examination and cardiac ultrasound examination were performed within 3 months before and after right heart catheterization;
2. mPAP > 25mmHg and PVR< 3woods (measured by right heart catheter) and pulmonary vascular resistance was collected as PAH group whereas Healthy Volunteers as non-PAH control group in developement corhort;
3. sPAP > 36mmHg (measured by echocardiography) was collected in validation corhort.

Exclusion Criteria:

1.Cancer; 2. The quality of chest CT and cardiac ultrasound images is poor; 3.Pulmonary vascular segmentation is affected by thoracic organ displacement or pulmonary vascular complete occlusion due to diseases ,such as spinal deformity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The development cohort is case_control research, composed of patients diagnosed with PAH and healthy control group from 2018.10 to now in RenjiH and Jiangsu Province Hospital.
  The validation cohort is prospective study to test the accuracy of diagonisis model, composed of patients are suspected as PAH or healthy volunteer by echocardiography form other medical institutions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
DIAGONOSIS | 1 year
  The patient is diagnosed PAH or not by right heart catheter

CONTACTS AND LOCATIONS:
Overall Officials: Jieyan Shen, PhD, Study Chair — Shanghai Jiao Tong University School of Medicine Affiliated Renji Hospital
Locations (1):
- Renji Hospital, Shanghai, China

REFERENCES:
- [Derived] Wan C, Chen M, Tong J, Wang A, Ruan B, Shen J. Prognostic effect of left ventricular-pulmonary arterial coupling indicator in pulmonary arterial hypertension. Int J Cardiol. 2025 Sep 1;434:133347. doi: 10.1016/j.ijcard.2025.133347. Epub 2025 May 1. PMID 40318737